CLINICAL TRIAL: NCT05660174
Title: Identification of Preoperative Parameters to Predict Acute Kidney Injury Risk Following Vascular or Digestive Surgery
Acronym: SCOPING
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/699
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Acute Kidney Injury
Keywords: Vascular Surgical Procedures; Digestive surgery; Vascular surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with a digestive surgery procedure
- Patient with a vascular surgery procedure

SUMMARY:
The study aims to identify the preoperative parameters associated with the risk of postoperative acute kidney injury (in particular the parameters of the SPARK score) in patients of the Besançon University Hospital who have undergone digestive or vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Digestive surgery or vascular surgery at Besancon University Hospital between 01/01/2019 and 31/12/2019 (retrospective) or between 01/01/2023 and 31/12/2023 (prospective)

Exclusion Criteria:

* No preoperative creatinine value
* Outpatient surgery
* Surgery other than digestive or vascular (organ procurement surgery/nephrectomy surgery/renal transplantation)
* Kidney/urinary tract surgery
* Arteriovenous fistula surgery
* End-stage renal disease or renal replacement therapy, except for renal transplant patients
* Acute kidney injury KDIGO≥1 within 2 weeks before surgery
* Patients in need of emergency surgery for ongoing haemorrhage
* Legal incapacity or limited legal capacity
* Subjects with no social security coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a digestive or vascular surgery procedure between 01/01/2019 and 01/06/2021 (retrospective) or between 01/01/2023 and 31/12/2023 (prospective), at the University Hospital of Besançon
Sampling Method: Probability Sample
Enrollment: 2626 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of acute kidney injury | 2 weeks after surgery
  Occurrence of acute kidney injury within 2 weeks after surgery, as defined by the 2012 KDIGO (Kidney Disease: Improving Global Outcomes) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Courivaud, Prof., Principal Investigator — Centre Hospitalier Universitaire de Besançon
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No